CLINICAL TRIAL: NCT07054671
Title: Investigating the Effects of Elderberry-Based Functional Beverage on Exercise Performance, Muscle Structure, and Gut-Muscle Axis: A Randomized Controlled Intervention Trial
Brief Title: Effects of an Elderberry-Based Functional Beverage on Exercise Performance, Muscle Structure, and the Gut-Muscle Axis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Gul Akduman, Research Assistant, Department of Nutrition and Dietetics, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MAKU-AKDUMAN-3501-2025
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Exercise; Anthocyanins; Muscle Size
Keywords: Anthocyanins; Exercise; Functional food; Muscle strength; Microbiota
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderberry Beverage Group (Experimental): Participants will consume an anthocyanin-rich elderberry-based functional beverage daily for 12 weeks while following a combined exercise protocol (2 days resistance + 1 day endurance training per week).
  Intervention;
  * Dietary Supplement (Elderberry-Based Functional Beverage)
  * A polyphenol and anthocyanin-rich beverage formulated from Sambucus nigra L., consumed once daily.
  Interventions: Dietary Supplement: Elderberry-Based Functional Beverage
- Placebo Beverage Group (Placebo Comparator): Participants will consume a placebo beverage that is matched in color and taste but does not contain polyphenols or anthocyanins, while following the same combined exercise protocol.
  Intervention:
  * Type: Placebo (Placebo Beverage)
  * A non-bioactive beverage matched for flavor and appearance, consumed once daily.
  Interventions: Dietary Supplement: Placebo Beverage

INTERVENTIONS:
Dietary Supplement: Elderberry-Based Functional Beverage — A polyphenol- and anthocyanin-rich beverage derived from Sambucus nigra L., administered once daily for 12 weeks as a dietary supplement.
  Other Names: 1
  Arms: Elderberry Beverage Group
Dietary Supplement: Placebo Beverage — A placebo beverage that mimics the elderberry drink in color and flavor but contains no polyphenols or bioactive compounds. Consumed once daily for 12 weeks.
  Arms: Placebo Beverage Group

SUMMARY:
Introduction: Increasing sedentary lifestyle, microbiota imbalance and exercise-induced muscle fatigue are among the main causes of metabolic stress and performance decline, even in young individuals. The potential effects of functional foods-particularly polyphenol and anthocyanin-rich beverages-on both gut microbiota and muscle performance have attracted attention in recent years. In this context, intervention studies focused on the gut-muscle axis represent a promising and valuable area of research.

Objective: This study aims to investigate the effects of a functional beverage enriched with anthocyanins and polyphenols -extracted from Sambucus nigra L. (black elderberry)- combined with a regular exercise program on muscle performance, muscle morphology, fatigue level, and gut microbiota composition in healthy individuals.

Method: This 12-week double-blind, randomized, placebo-controlled trial will include participants adhering to a berry-free diet. Participants will be randomly assigned to two groups: the intervention group will consume a functional elderberry beverage formulated with high-purity anthocyanins obtained via supercritical CO₂ extraction; the control group will receive a placebo beverage with matched taste and energy content but without active compounds. Both groups will engage in a structured combined exercise program (3 days/week). Pre- and post-intervention assessments will include gut microbiota profiling (16S rRNA sequencing), short-chain fatty acid analysis, systemic biomarkers, muscle morphology (via ultrasound), exercise performance, and body composition. Mediator analyses will be used to explore the role of the gut-muscle axis in the observed effects.

Unique value: This project represents one of the few human-based intervention studies systematically evaluating the interaction between functional beverages, exercise, and microbiota through the lens of muscle fiber-type-specific adaptations. Furthermore, by integrating mediator analyses and multi-level outcome measures, the study aims to elucidate the physiological relevance of the gut-muscle axis in a holistic manner. The development, standardization, and sensory evaluation of the elderberry-based beverage also contribute valuable insights to functional product innovation.

DETAILED DESCRIPTION:
In modern times, the increasing prevalence of sedentary lifestyles, age-related decline in muscle function, and gut dysbiosis have been shown to negatively affect both metabolic health and muscular performance. These problems are not only observed in the elderly population but also in physically active young individuals, manifesting as exercise-induced fatigue, reduced performance, and impaired immune function. Sustaining muscle performance is closely related not only to physical fitness but also to maintaining gut microbiota balance and controlling inflammation.

The health effects of functional foods have become a focal point in multidisciplinary research in recent years. In this context, developing functional beverages rich in bioactive compounds such as polyphenols, flavonoids, and anthocyanins offers new research opportunities, particularly in the fields of exercise physiology and immune response. This study aims to evaluate the effects of an anthocyanin-enriched functional beverage derived from Sambucus nigra L. (elderberry) on muscle performance, fatigue, and the gut-muscle axis in healthy individuals participating in a combined exercise protocol.

Elderberry is a bioactive source noted for its high anthocyanin content, showing antioxidant and anti-inflammatory effects, and its potential to positively modulate gut microbiota. Since anthocyanins are only minimally absorbed in the small intestine, a large proportion reaches the colon, where they are fermented by the gut microbiota into various phenolic acids. This fermentation process may support the proliferation of beneficial species such as Bifidobacterium and Lactobacillus, while reducing pathogenic species such as Clostridium perfringens. Furthermore, elderberry polyphenols may promote the growth of anti-inflammatory species like Akkermansia muciniphila and Faecalibacterium prausnitzii. These microbial changes-especially the increase in short-chain fatty acids (SCFAs), particularly butyrate-have been associated with improved immune response, gut barrier integrity, and muscle metabolism. In vivo studies have shown that anthocyanin supplementation enhances microbial diversity and stimulates SCFA production, thereby helping to suppress inflammation. Within the so-called "gut-muscle axis," SCFAs-especially butyrate-play roles in muscle protein synthesis, mitochondrial function, and inflammation regulation. Some animal studies have also shown that modulation of microbiota composition via probiotics and polyphenol supplementation positively affects muscle mass and endurance.

Therefore, the researchers hypothesize that the elderberry-based beverage may reduce exercise-induced muscle fatigue and enhance performance not only through systemic antioxidant mechanisms but also by regulating gut microbiota. Consequently, this study will also assess how the microbiota changes induced by the beverage affect muscle metabolism.

A combined exercise protocol (2 days of resistance + 1 day of endurance) has been chosen, as it is an effective model for stimulating both cardiorespiratory capacity and muscle function. The literature highlights that endurance training improves mitochondrial biogenesis, oxidative capacity, and lactate clearance, whereas resistance training increases muscular strength and hypertrophy. It has been demonstrated that combined protocols are more effective for improving metabolic health and functional capacity.

To evaluate not only general muscle hypertrophy but also fiber-type-specific physiological adaptations, three muscle groups will be assessed: quadriceps, soleus (Type I fiber dominant), and gastrocnemius (Type II fiber dominant). These muscles were selected based on their well-defined morphological and metabolic profiles in the literature, allowing for indirect assessment of anthocyanins and polyphenols on mitochondrial function and oxidative stress. This makes the study one of the few human-based interventions that systematically investigates the effects of functional foods on exercise physiology with a muscle fiber-type-specific approach.

This study is among the few examples in the literature that evaluate functional beverages not only at the bioactive compound level but also in the context of exercise physiology and microbiota interaction. Most current research focuses on the short-term effects of polyphenol supplementation or isolated microbiota outcomes. However, this project aims to evaluate the holistic effects of a polyphenol/anthocyanin-rich functional beverage on both performance physiology and gut microbiota. Furthermore, the mediating role of the gut-muscle axis will be explored through quantitative measurements. This approach introduces a new methodological framework for both bioactive food development and microbiota-based exercise science. To date, there has been no human-based randomized controlled trial combining exercise, microbiota, and functional beverage interventions in the same design.

ELIGIBILITY:
Inclusion Criteria:

* Engaging in regular physical activity at least 2 days per week
* Body Mass Index (BMI) between 18.5 and 29.9 kg/m²
* No use of antibiotics, probiotics, or prebiotics within the past 3 months
* No history of chronic illness or autoimmune disorders
* Physically able and eligible to participate in exercise training
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Known food allergies
* Regular use of medications such as corticosteroids, NSAIDs, or immunosuppressants
* Professional-level athletes
* All participants will be instructed to avoid consuming any products containing berries (fresh, frozen, dried, jam, juice, or supplements) during the intervention period. A "berry-free diet" will be implemented as part of the study protocol. At baseline, a short Food Frequency Questionnaire (FFQ) will be administered to assess participants' berry consumption habits over the past month. The FFQ will include 10 commonly consumed berries in Türkiye: strawberry, raspberry, blackberry, blueberry, elderberry, mulberry, redcurrant, blackcurrant, aronia, and goji berry. Each item will be scored on a scale from 0 (never) to 4 (daily), and the total score will represent the individual's berry consumption score. Participants with a total baseline score of ≥10 will be excluded to minimize confounding from prior polyphenol exposure. The FFQ will only be used to assess baseline habits and ensure compliance with the berry-free protocol; it will not be used in primary outcome analyses.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Muscle Fatigue (VAS Score) After 12 Weeks | Baseline and Week 12
  Muscle fatigue perception will be assessed using a 10-point visual analog scale (VAS), where 0 indicates no fatigue and 10 indicates extreme fatigue.
  Unit of Measure: Units on a 10-point scale Interpretation: A lower score indicates improvement.
Change in Time-to-Exhaustion Performance After 12 Weeks | Baseline and Week 12
  Muscle endurance will be assessed by measuring the time (in seconds) a participant can continue a standardized exercise until exhaustion.
  Unit of Measure: Seconds Interpretation: A higher time indicates improvement.

SECONDARY OUTCOMES:
Change in Gut Microbiota Composition | Baseline and Week 12
  Fecal samples will be collected to evaluate taxonomic and functional changes in gut microbiota using 16S rRNA sequencing. Relative abundance of key microbial taxa (e.g., Akkermansia muciniphila, Faecalibacterium prausnitzii) and alpha diversity indexes will be reported.
  Unit of Measure: Alpha diversity index units (e.g., Shannon index); relative abundance (%) Interpretation: Increased diversity or beneficial taxa indicate improvement
Change in Muscle Architecture Parameters | Baseline and Week 12
  Muscle architecture will be assessed via ultrasound by measuring muscle thickness (mm) and pennation angle (degrees) separately for each muscle. Each parameter will be reported individually.
  Unit of Measure: millimeters (mm) and degrees (°) Interpretation: Increases in muscle thickness and pennation angle reflect hypertrophic adaptations.
Change in Exercise Performance (VO₂peak) | Baseline and Week 12
  Maximal oxygen consumption (VO₂peak) will be measured using a graded treadmill test following standard protocols. Improved values will reflect enhanced aerobic capacity.
  Unit of Measure: mL/kg/min Interpretation: Higher VO₂peak indicates improved aerobic performance.

CONTACTS AND LOCATIONS:
Locations (1):
- MAKU Department of Nutrition and Dietetics, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) will depend on the ethical committee's final approval and data protection considerations. If permitted, de-identified data may be shared with qualified researchers upon reasonable request following publication. Until ethical clearance for data sharing is obtained, no commitment can be made.